CLINICAL TRIAL: NCT07311746
Title: Phase Ib/II Trial of Cladribine/Ruxolitinib/Venetoclax in Patients With Relapsed/Refractory T-cell Prolymphocytic Leukemia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1464; NCI-2025-09671 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-12-29; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: T-cell Prolymphocytic Leukemia; Refractory T-Cell Prolymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Prolymphocytic, T-Cell | interventions — ruxolitinib; Cladribine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SingleArm: Phase 1b/II - ESC/EXP Treatment with Ruxolitinib + Cladribine + Venetoclax (Experimental): Participants will receive treatment on an inpatient basis for the first cycle and can be administered on an outpatient basis for the subsequent cycles.
  Interventions: Drug: Ruxolitinib; Drug: Cladribine; Drug: Venetoclax

INTERVENTIONS:
Drug: Ruxolitinib — Given orally
  Other Names: Jakafi
Drug: Cladribine — Given by injection
  Other Names: Mavenclad
Drug: Venetoclax — Taken by mouth
  Other Names: Venclexta

SUMMARY:
The goal of this clinical research study is to learn if the combination of ruxolitinib with cladribine and venetoclax can help to control the disease in patients with R/R T-PLL.

DETAILED DESCRIPTION:
Primary Objective:

• To evaluate the safety and tolerability of Ruxolitinib in combination with Cladribine and Venetoclax in patients with R/R T-PLL.

Secondary Objectives:

* To evaluate the EFS in patients with T-PLL treated with Ruxolitinib in combination with Cladribine and Venetoclax.
* To evaluate response (CR, including CRi, or PR) of Ruxolitinib in combination with Cladribine and Venetoclax in patients with T-PLL.
* To assess the time to response, response duration, and OS in patients with T-PLL treated with Ruxolitinib in combination with Cladribine and Venetoclax.

Exploratory Objective:

• To explore correlation of genomic profile, baseline patient and disease characteristics, and response to BCL-2 inhibition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed a diagnosis T-PLL that is relapsed or refractory after prior treatment.
2. Age ≥ 18 years.

   * Patients must not have had T-PLL directed chemotherapy or antibody therapy for 7 days prior to starting ruxolitinib. However, patients with rapidly proliferative disease may receive hydroxyurea or decadron until 24 hours prior to starting therapy on this protocol.
   * Patients with a prior or concurrent malignancy whose natural history or treatment does not interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
3. Adequate organ function as defined below:

   * liver function (bilirubin < 2mg/dL, AST and ALT <3 x ULN - or ≤5 x ULN if related to leukemic involvement);
   * kidney function (estimated creatinine clearance > 50);
   * known cardiac ejection fraction of ≥ 45% within the past 3 months prior to enrolling on the trial;
   * Platelet count of ≥ 30,000 (unless determined to be due to disease involvement).
4. ECOG performance status of ≤ 2.
5. For patients with evidence of chronic HBV infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
6. Patients with a history of HCV infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
7. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.

   The effects of ruxolutinib on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:
   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure.
8. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), IUD, Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
9. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ruxolitinib and venetoclax administration.
10. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.

Exclusion Criteria:

1. Pregnant women are excluded from this study because the agent used has the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided.
2. Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, clinically significant or cardiac arrhythmia
3. Patient with documented hypersensitivity to any of the components of the therapy program.
4. Patients with known active, uncontrolled CNS leukemia will not be eligible.
5. Patients with prior treatment with a JAK1, JAK2, or JAK3 inhibitor will not be eligible.
6. Men and women of childbearing potential who do not practice contraception.
7. Known history of active HIV infection (HIV 1/2 antibodies).
8. Active HBV or HCV infection that requires treatment or at risk for HBV reactivation.

   Hepatitis B virus DNA and HCV RNA must be undetectable upon testing. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Prior test results obtained as part of standard of care that confirm a subject is immune and not at risk for reactivation (ie, hepatitis B surface antigen negative, surface antibody positive) may be used for purposes of eligibility and tests do not need to be repeated. Subjects with prior positive serology results must have negative polymerase chain reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.
9. Patients who are receiving any other investigational agents.
10. Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Kadia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org